CLINICAL TRIAL: NCT07356180
Title: Epigenetic Regulation of Physically Active Lifestyle on Placental Development
Brief Title: Physical Acvitiy in Pregnancy
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Jun Seok Son, Assistant Professor, University of Maryland, Baltimore
Other Study IDs: HP-00099879
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Pregnant Women; Gestational Diabetes; Obese But Otherwise Healthy Participants; Overweight (BMI > 25); Gestational Diabetes Mellitus in Pregnancy
Keywords: maternal exercise; gestational diabetes; maternal physical activity; pregnancy; placental function; fetal development; maternal obesity; observational study; placental mitochondria; lifestyle intervention; pregnancy outcomes
MeSH Terms: conditions — Diabetes, Gestational; Overweight; Pregnancy in Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples With DNA — Biospecimens collected during pregnancy and at delivery will be retained for analysis of placental function, including potential DNA extraction for research purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Con: pre-pregnancy BMI 18.5-24.9, no gestational diabetes
  Interventions: Behavioral: Pregnancy Physical Activity Questionnaire (PPAQ)
- overweight/obesity group: pre-pregnancy BMI of 25 or greater, no gestational diabetes
  Interventions: Behavioral: Pregnancy Physical Activity Questionnaire (PPAQ)
- Gestational DM group: pre-pregnancy BMI 18.5-24.9 with gestational diabetes
  Interventions: Behavioral: Pregnancy Physical Activity Questionnaire (PPAQ)
- gestational DM + overweight/obesity group: pre-pregnancy BMI of 25 or greater, with gestational diabetes
  Interventions: Behavioral: Pregnancy Physical Activity Questionnaire (PPAQ)

INTERVENTIONS:
Behavioral: Pregnancy Physical Activity Questionnaire (PPAQ) — The PPAQ is a semiquantitative questionnaire that asks respondents to report the time spent participating in 32 activities including household/caregiving (13 activities),occupational (5 activities), sports/exercise (8 activities), transportation (3 activities), and inactivity (3 activities).
  For each activity, respondents are asked to select the category that best approximates the amount of time spent in that activity per day or week during the currenttrimester. Possible durations range from 0 to 6 or more hours per day and from 0 to 3 or more hours per week.

SUMMARY:
The goal of this observational study is to learn how a physically active lifestyle during pregnancy affects placental development and function. The main question it aims to answer is:

Does regular physical activity during pregnancy improve placental function and support healthy fetal growth?

Pregnant participants will provide biological samples and health information during pregnancy and at delivery. The study will use these samples to examine how activity levels relate to placental energy production and overall health.

DETAILED DESCRIPTION:
This observational study aims to examine how a physically active lifestyle during pregnancy affects placental function and fetal development. We will enroll pregnant participants and collect biological samples, including blood and placental tissue after delivery. The study will measure markers of placental energy production and other indicators of placental health to understand the mechanisms by which maternal physical activity may influence fetal growth.

Data collected will also include health information, lifestyle questionnaires, and activity assessments during pregnancy. Participants will not need to change their normal exercise habits. The results of this study may help identify how maternal physical activity supports placental and fetal health, which could inform future recommendations for healthy pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female and their newborn infant(s)
* Aged 18-45 (pregnant female), age 0-60 days of life (newborn infant)
* English speaking
* Screened for gestational diabetes with standard glucose tolerance test between 24w - 41w gestation
* Delivered at gestational age 34week-41weeks
* Delivered via non-emergent Cesarean section during weekday hours
* No known infectious disease (ex: HIV, HepC)

Exclusion Criteria:

* Women <18yo or >45yo
* Non-English speaking
* Pre-existing diabetes or diagnosed with diabetes prior to 24weeks
* Required complex diets/supplements not related to the pregnancy (i.e. malnutrition)
* Known severe fetal anomalies or genetic disorder
* Placenta accreta spectrum
* Emergent cesarean delivery performed due to fetal distress
* Known infectious disease (ex: HIV, HepC)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of pregnant individuals receiving prenatal care and/or delivering at affiliated clinical sites of the University of Maryland, Baltimore and surrounding community healthcare settings. Participants will be recruited from local obstetric clinics and hospital-based prenatal care programs. The study represents a community-based sample of pregnant individuals with varying levels of physical activity during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Placental mitochondrial function | At delivery
  Placental mitochondrial function will be assessed using markers of mitochondrial biogenesis and energy metabolism measured in placental tissue collected at delivery. Outcomes will be examined in relation to maternal physical activity levels during pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical System, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Results of our study will not be shared with the subjects. We plan on publishing our results in a peer reviewed journal. We also plan to present the results as a thesis dissertation for Dr. Esteves. We also hope the results will generate evidence for benefits of physical activity during pregnancy, which will lead to seeking extramural NIH grants for cohort study of pregnant women with exercise programs.